CLINICAL TRIAL: NCT04948658
Title: Gonadal Tissue Freezing for Fertility Preservation in Individuals at Risk for Ovarian Dysfunction, Premature Ovarian Insufficiency and Clinically Indicated Gonadectomy
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000106; 000106-CH
Record Dates: First submitted 2021-07-01; First posted 2021-07-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Turner Syndrome; Post-menarcheal Adolescents; Ovarian Disfunction; Galactosemia; Variations in Sex Characteristics; Differences in Sex Development
Keywords: OVARIAN FUNCTION; Natural History; follicle loss; Variations in Sex Characteristics; Differences in Sex Development
MeSH Terms: conditions — Turner Syndrome; Galactosemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Adolescents with DOR: Adolescents with diminished ovarian reserve (DOR) who respond poorly to ovarian stimulation for egg freezing.
- Adolescents with POI: Adolescent females up to age 21 years old, who have undergone menarche and are subsequently diagnosed with POI and their last menstrual period occurred within 2 years of presentation.
- Individuals receiving high-risk gonadotoxic therapy: Individuals (2-35 years) receiving high-risk gonadotoxic therapy at the NIH Clinical Center who are at high risk for developing premature ovarian insufficiency and infertility.
- Individuals with variations in sex characteristics (or differences in sex development, DSD): Individuals with variations in sex characteristics (or differences in sex development, DSD) who undergo gonadectomy for clinical indications.
- Turner Syndrome and galactosemia: Individuals with Turner Syndrome prior to menarche aged 2 years to 12 years, who have not previously demonstrated signs of premature ovarian insufficiency (FSH>25 IU/L).
- Turner Syndrome with Y material: Children and adolescents who have Turner syndrome with Y material and undergo prophylactic gonadectomy.

SUMMARY:
Background:

Turner Syndrome, galactosemia, and premature ovarian insufficiency are all conditions that may make it very hard or impossible for a person to become pregnant and have their own child. Researchers want to learn more about why this happens and if freezing Gonadal tissue allows for fertility preservation.

Objective:

To find out why people with certain conditions have can have premature ovarian insufficiency (POI or early menopause) and individuals with variations in sex characteristics have trouble getting pregnant and if freezing the gonads tissue from them will help to have their own child in the future.

Eligibility:

Individuals aged 2-21 who have Turner Syndrome or galactosemia. Also, females aged 13-21 with premature ovarian insufficiency, individuals with variations in sex characteristics, and individuals 2-35 receiving high-risk gonadotoxic therapy

Design:

Participants will be screened with a medical history.

Participants may have a physical exam and blood tests. Their body measurements may be taken. These include weight, height, arm span, skin fold, and sitting height. They may fill out surveys about their quality of life, body image, and health.

Participants may have a transabdominal pelvic ultrasound. A probe will be placed on their belly and will take pictures of the organs in the pelvis. They may have a transvaginal pelvic ultrasound performed while asleep in the operating room if needed.

Participants may have surgery to remove an gonads and skin biopsy. The removed tissue will be frozen and stored. The tissue will have to be stored for many years. NIH will pay to store the tissue for 1 year. After that, participants will have to pay for storage.

A piece of the gonads (no more than 20%) will be used for research

Travel, lodging and meals for participants traveling greater than 50 miles will be reimbursed based off the government rate. Local participants will not be reimbursed.

Participants will have a checkup 6 weeks after surgery one or more follow-up visits 6-18 months after surgery. They may have phone follow-up every 12-24 months after surgery.

Participation will last 30 years.

DETAILED DESCRIPTION:
Study Description:

Gonadal tissue cryopreservation will be evaluated in individuals with Turner Syndrome, galactosemia, post-menarcheal adolescents with recent premature ovarian insufficiency, and children/adolescents conditions associated with POI and with diminished ovarian reserve (DOR) who have contraindication to ovarian stimulation as well as those with diminished ovarian reserve who did not respond to ovarian stimulation, and individuals with variations in sex characteristics (VSD or differences in sex development, DSD) including those with Turner syndrome with Y chromosome material and those with conditions that require high risk gonadotoxic therapy.

Objectives:

Primary Objectives: After initial evaluation of number and quality of follicles/gametes, the remaining tissue will be utilized to perform research regarding mechanisms of follicle/gametes loss in the included conditions.

a. We will perform next generation sequencing on the tissue collected from study participants and ovaries from cadaveric organ donors on cardiopulmonary support. Additionally, some ovarian tissue from patients undergoing gonadotoxic therapy will function as controls.

Hypothesis: next generation sequencing from tissue obtained from gonads in individuals with these conditions will differ significantly from that of controls. Such differences may allow for further hypothesis development regarding the underlying mechanism of follicle loss and/or dysfunction in individuals with these conditions.

Secondary Objective: This protocol is designed to evaluate the feasibility (meaning a reasonable expectation of future fertility based on the anatomy, histology, and physiology of fresh gonadal tissue as well as the effects after freezing and thawing) of gonadal tissue cryopreservation (GTC) for fertility preservation in children with increased risk of loss of gonadal function due to underlying genetic conditions including Turner syndrome or galactosemia and post-menarcheal adolescents with a recent development of premature ovarian insufficiency (POI) or children/adolescents with conditions associated with POI and presenting with diminished ovarian reserve (based on laboratory findings of low AMH (<1.0 ng/mL) and/or mildly elevated FSH (>10 U/L) or those who do not respond to ovarian stimulation for oocyte cryopreservation due to lower follicle counts) or individuals with variations in sex characteristics.

1. The feasibility GTC as a fertility preservation option in these individuals will be evaluated through evaluation of number and quality of follicles/gametes found in the tissue prior to freezing and after thawing.
2. Lack of follicles/gametes in the gonadal tissue will confirm that GTC is not a viable option for fertility preservation for these populations.
3. An attempt to correlate laboratory and imaging markers with follicle/gamete presence and number will be made.

b. Hypothesis: Young individuals with Turner syndrome, variations of sex characteristics, classic galactosemia and adolescents with recent POI, and children/adolescents with underlying conditions associated with POI presenting with DOR harbor populations of follicles/gametes which may be preserved through gonadal tissue cryopreservation for future fertility. There will be a variety of follicular findings which will correlate with patient s anti-Mullerian hormone (AMH), age and underlying condition.

c. Depending on their underlying condition, individuals with VSC will have gametes (follicles and/or spermatogonia).

d. Loss of follicles with cryopreservation and thawing will be similar to that of non-affected individuals.

Tertiary Objectives:

Research regarding inhibition and activation of follicles within the tissue will be undertaken.

1. Tissue will be treated with known inhibitors and activators and next generation sequencing will be performed in order to assess gene expression before and after treatment.
2. To create a national database of human ovarian tissue of individuals who are undergoing OTC in order to elucidate short and long term outcomes including complication and reproductive health parameters.

Hypothesis: Primordial follicles within gonadal tissue in individuals with these conditions may be inhibited from activating. Such techniques may allow for a decrease in follicle loss with freezing and thawing as well as possible future development of novel treatments to prevent accelerated follicle loss in individuals and adolescent affected by these conditions. Promoting follicle activation prior to re-implantation of the tissue may improve the possibility of achieving pregnancy after tissue re-implantation

Endpoints:

Primary Endpoints:

1. Tissue for research: Next generation sequencing will be performed on tissues of affected individuals and compared to age matched controls: patients who undergo GTC for solid organ tumors far from the reproductive system or cadaveric organ donors on cardiopulmonary support. This will allow for specific cellular type comparisons within the ovary and exploratory research regarding possible mechanisms of follicle loss in these populations.
2. Next generation sequencing on fresh compared to frozen and thawed tissue. This will assess what transcription changed occur due to the freezing process.

Secondary Endpoint:

1. Evaluation of density and quality of follicles/gametes in the gonads of individuals with increased risk of loss of gonadal function due to underlying genetic conditions including Turner syndrome or galactosemia and post-menarcheal adolescents with a recent development of premature ovarian insufficiency (POI) or children/adolescents with conditions associated with POI and presenting with diminished ovarian reserve (based on laboratory findings of low AMH (<1.1 ng/mL) and mildly elevated FSH (10-25 U/L) or those who do not respond to ovarian stimulation for oocyte cryopreservation due to lower follicle counts) or individuals with variations in sex characteristics.
2. Correlation of follicle/gamete density and quality with markers such as age, AMH, condition.
3. Comparison of hormone levels such as AMH, FSH, LH, and Estradiol between patients and controls.
4. Long term data regarding surgical complications

Tertiary Endpoint:

-Evaluate changes in single next generation sequencing in tissue before and after treatment with primordial follicle inhibitors and activators. The remaining tissue will be cryopreserved for future experiments.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

-Individuals with Turner Syndrome prior to menarche aged 2 years to 12 years whose families seek to store ovarian tissue for possible future use.

Or

Individuals with galactosemia (age 2-21)

Or

Adolescent females up to age 21 years old, who have undergone menarche and are subsequently diagnosed with premature ovarian insufficiency and their last menstrual period occurred within 2 years of presentation. Diagnosis of POI is based on 2 elevated FSH concentrations obtained over 1 month apart.

Or

Children or adolescents who have diminished ovarian reserve based on laboratory findings or who respond poorly to ovarian stimulation for egg freezing.

Or

Individuals with variations in sex characteristics (or differences in sex development, DSD) including Turner syndrome with Y chromosome material who undergo prophylactic gonadectomy for clinical indications.

Or

Individuals (2-35 years) receiving high-risk gonadotoxic therapy at the NIH Clinical Center who are at high risk for developing premature ovarian insufficiency and infertility.

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability of subject, parents, or guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Individuals older than 7 years with psychological, psychiatric, or other conditions which prevent giving fully informed consent or assent.
* Individuals with a pelvic mass tumor noted on pre-operative ultrasound, will undergo usual care for the underlying condition and will not undergo oophorectomy for ovarian tissue cryopreservation.
* Individuals whose underlying medical condition significantly increases their risk of complications from anesthesia and surgery.
* Females with POI due to chemotherapy or radiation treatment
* Pregnancy or lactation
* Individuals with VSC who choose to retain gonads after clinical consulting.
* Individuals with Turner Syndrome who have an undetectable AMH based on testing laboratory reference range.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with Turner Syndrome prior to menarche aged 2 years to 12 years, who have not previously demonstrated signs of premature ovarian insufficiency (FSH>25 IU/L) and have detectable anti-Mullerian hormone (AMH). Individuals with classic galactosemia age 2-21. Individuals with Turner Syndrome with Y chromosome material who undergo prophylactic gonadectomy. Adolescent females aged 13 to 21 years old who have undergone menarche and are subsequently diagnosed with premature ovarian insufficiency with their last menstrual period having occurred within 2 years of presentation. Children and Adolescents (2-21) with diminished ovarian reserve who have contraindication to ovarian stimulation as well as those with diminished ovarian reserve who did not respond to ovarian stimulation. Individuals with variations in sex characteristics (or differences in sex development, DSD) who undergo gonadectomy for clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Single cell/nucleus RNA sequencing | before and after cryopreservation
  Single cell/nucleus RNA sequencing on fresh compared to frozen and thawed tissue. This will assess what transcription changed occur due to the freezing process.
Tissue for research | before and after cryopreservation
  initial evaluation of number and quality of follicles before and after cryopreservation

SECONDARY OUTCOMES:
Evaluate gonadal tissue | before and after cryopreservation
  The ability to safely offer a fertility preservation option to individuals who are at high risk such as POI, DOR and VSC.
Evaluate changes in single cell/nucleus RNA sequencing | before and after cryopreservation
  Evaluate changes in single cell/nucleus RNA sequencing in tissue before and after treatment with primordial follicle inhibitors and activators.
Compare hormone levels | before and after cryopreservation
  Comparison of hormone levels such as AMH, FSH, LH, and Estradiol between patients and controls.
density and quality of follicles in the ovaries | before and after cryopreservation
  Evaluation of density and quality of follicles in the ovaries of girls with Turner syndrome, galactosemia and post-menarcheal adolescent with premature ovarian insufficiency before and after cryopreservation and thawing
Correlation of follicle density and quality with markers such as age, AMH, condition. | before and after cryopreservation
  Correlation of follicle density and quality with markers such as age, AMH, condition.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are trying to figure out if we want to share IPD.

REFERENCES:
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org. Fertility preservation and reproduction in patients facing gonadotoxic therapies: an Ethics Committee opinion. Fertil Steril. 2018 Aug;110(3):380-386. doi: 10.1016/j.fertnstert.2018.05.034. PMID 30098684
- [Background] Martinez F; International Society for Fertility Preservation-ESHRE-ASRM Expert Working Group. Update on fertility preservation from the Barcelona International Society for Fertility Preservation-ESHRE-ASRM 2015 expert meeting: indications, results and future perspectives. Fertil Steril. 2017 Sep;108(3):407-415.e11. doi: 10.1016/j.fertnstert.2017.05.024. Epub 2017 Jul 21. PMID 28739117
- [Background] Andersen ST, Pors SE, Poulsen LC, Colmorn LB, Macklon KT, Ernst E, Humaidan P, Andersen CY, Kristensen SG. Ovarian stimulation and assisted reproductive technology outcomes in women transplanted with cryopreserved ovarian tissue: a systematic review. Fertil Steril. 2019 Nov;112(5):908-921. doi: 10.1016/j.fertnstert.2019.07.008. Epub 2019 Oct 6. PMID 31594631
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000106-CH.html